CLINICAL TRIAL: NCT02751827
Title: Predicting Severe Toxicity of Targeted Therapies in Elderly Patients With Cancer
Acronym: PreToxE
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Agence Nationale de sécurité du Médicament (Other)
Responsible Party: Sponsor
Other Study IDs: IB 2015-02
Record Dates: First submitted 2016-04-25; First posted 2016-04-26 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2021-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One blood sample before treatment initiation (Cycle 1 Day predose) for pharmacogenomics.
  One blood sample at the end of the firth month of treatment (postdose) for pharmacokinetic
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prospective cohort: Prospective cohort involving patients treated in four distinct centers. Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
  All patients without major violations of the eligibility criteria are included in the eligible population. In case of violation of the eligibility criteria, the steering committee will assess for each patient, whether the violation is minor or major.
  All eligible patients who have received at least one TKI administration were included in analysis.
  Interventions: Other: Blood sample
- Retrospective cohort A: Retrospective cohort of patients treated at the Institut Bergonié (Bordeaux, France). Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
  All patients without major violations of the eligibility criteria are included in the eligible population. In case of violation of the eligibility criteria, the steering committee will assess for each patient, whether the violation is minor or major.
  All eligible patients who have received at least one TKI administration were included in analysis.
- Retrospective cohort B: Retrospective cohort of patients treated at the Centre Antoine Lacassagne(Nice, France). Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
  All patients without major violations of the eligibility criteria are included in the eligible population. In case of violation of the eligibility criteria, the steering committee will assess for each patient, whether the violation is minor or major.
  All eligible patients who have received at least one TKI administration were included in analysis.

INTERVENTIONS:
Other: Blood sample — One blood sample before treatment initiation (Cycle 1 Day predose) for pharmacogenomics
  One blood sample at the end of the firth month of treatment (postdose) for pharmacokinetic
  Groups: Prospective cohort

SUMMARY:
In order to assess the important issue of the safety of antiangiogenic TKI in geriatric population we set up this project which aims to identify, among clinical, biological, pharmacokinetic data, predictive factors for severe toxicity of antiangiogenic TKI (sunitinib, sorafenib, pazopanib, regorafenib, axitinib) in patients over 70 year-old.

DETAILED DESCRIPTION:
This is a prospective cohort with collection of biological samples, including 300 patients > 70 year-old treated in multicenter with antiangiogenic TKI regularly approved for metastatic cancers. Data on clinical and biological characteristics of the patient, disease and treatment as well as pharmacogenomics will be centrally collected at the beginning of the treatment. Drug exposure-safety analyses will be performed through assessment of drug through levels (Cmin). Primary endpoint is severe toxicity defined as treatment-related death, hospitalization or disruption of treatment for more than three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Treatment with pazopanib, regorafenib, sorafenib, sunitinib,axitinib in the context of market authorization
* Voluntary signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

* Patient treated in a context of clinical trial
* Patient with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients without major violations of the eligibility criteria are included in the eligible population. In case of violation of the eligibility criteria, the steering committee will assess for each patient, whether the violation is minor or major.
  All eligible patients who have received at least one TKI administration were included in analysis.
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebreton C, Cantarel C, Toulza E, Desgrippes R, Bozec L, Saada E, Ducoulombier A, Tardy M, Paillaud E, Lalet C, Bellera C, Italiano A. Incidence and prognostic factors of clinically meaningful toxicities of kinase inhibitors in older patients with cancer: The PreToxE study. J Geriatr Oncol. 2021 May;12(4):668-671. doi: 10.1016/j.jgo.2020.09.020. Epub 2020 Sep 23. PMID 32978101

RESULTS

PARTICIPANT FLOW:
Groups:
- Prospective Cohort: Prospective cohort involving patients treated in four distinct centers. Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
- Retrospective Cohort A: Retrospective cohort of patients treated at the Institut Bergonié (Bordeaux, France). Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
- Retrospective Cohort B: Retrospective cohort of patients treated at the Centre Antoine Lacassagne(Nice, France). Patients were treated with a tyrosine kinase inhibitor (TKI) prescribed as part of a marketing authorization (MA).
Period: Overall Study
Arm/Group | Prospective Cohort | Retrospective Cohort A | Retrospective Cohort B
Started | 41 | 171 | 100
Completed (Eligible and assessable population : All eligible patients who have received at least one TKI administration were included in analysis.) | 41 | 171 | 99
Not Completed | 0 | 0 | 1
Not completed — Only patient treated by TKI without anti-angiogenic action. He was excluded due to selection bias. | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and assessable population
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Cohort | Retrospective Cohort A | Retrospective Cohort B | Total
Number analyzed (Participants) | 41 | 171 | 99 | 311
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 79 [76 to 82] | 74 [72 to 78] | 76 [72 to 79] | 75 [72 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 98 | 36 | 150
  Male | 25 | 73 | 63 | 161
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 41 | 171 | 99 | 311

OUTCOME MEASURES:

1. Primary Outcome: Rate of Severe Toxicity
Description: Severe toxicity was defined as any TKI-related adverse events (AE) leading to any one of the following events: death, persistent or significant disability/incapacity (defined as a permanent physical or mental impairmentwhich seriously limits one or more functional capacities such as mobility, communication, self-care, self-direction, or interpersonal skills), unexpected hospitalization, drug discontinuation for more than three weeks or definitive discontinuation.
  All adverse events (AE) were graded as per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Time Frame: During treatment, up to 12 months or within 4 weeks following definitive treatment discontinuation, an average of 5 months.
Population: Eligible and assessable population : All eligible patients who have received at least one TKI administration were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Cohort | Retrospective Cohort A | Retrospective Cohort B
Number analyzed (Participants) | 41 | 171 | 99
Participants | 14 | 75 | 43

ADVERSE EVENTS:
Time Frame: During treatment, up to 12 months or within 4 weeks following definitive treatment discontinuation, an average of 5 months.
Description: All AE (all imputability) were collected, excepted for retrospectvie cohort B for which only treatment-related AE were collected.
  Following study protocol, SAE (i.e severe toxicity) were defined as any AE related to the treatment leading to any one of the following events: death, persistent or significant disability/incapacity, unexpected hospitalization, drug discontinuation for more than three weeks or definitive discontinuation. Hence, no SAE were unrelated to the treatment.
Arm/Group | Prospective Cohort | Retrospective Cohort A | Retrospective Cohort B
All-Cause Mortality (participants affected / at risk) | 21/41 | 62/171 | 46/99
Serious Adverse Events (participants affected / at risk) | 14/41 | 75/171 | 43/99
Other Adverse Events (participants affected / at risk) | 36/41 | 131/171 | 76/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Cohort (N=41) | Retrospective Cohort A (N=171) | Retrospective Cohort B (N=99)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Macrophage activation syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Digestive problems (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 26 (26) | 17 (18)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Deterioration of general condition (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cranial nerve infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 15 (15) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Tumor bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mood disorders (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective Cohort (N=41) | Retrospective Cohort A (N=171) | Retrospective Cohort B (N=99)
Anemia (Blood and lymphatic system disorders) | 6 (7) | 16 (16) | 11 (11)
Thrombopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3) | 11 (11)
Conjunctivitis (Eye disorders) | 0 (0) | 6 (6) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (6) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 16 (18) | 32 (32) | 30 (30)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 21 (21) | 15 (15)
Nausea (Gastrointestinal disorders) | 8 (8) | 6 (6) | 8 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 8 (8) | 1 (1)
Sphincter disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 10 (10) | 1 (1)
Fatigue (General disorders) | 27 (27) | 42 (42) | 56 (56)
Fever (General disorders) | 1 (1) | 4 (4) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Altered general condition (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 4 (4) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 16 (16) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 6 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 13 (13) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 3 (3) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 15 (15) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 5 (5) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 4 (4) | 3 (3)
Platelet count decreased (Investigations) | 7 (7) | 8 (8) | 10 (10)
Weight loss (Investigations) | 3 (3) | 4 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 16 (17) | 19 (19) | 25 (25)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 16 (16) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Severe undernutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Cramps (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 9 (10) | 9 (9) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Agueusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Vigilance disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 12 (12) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 6 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 7 (7) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 17 (17)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 26 (26) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythematous lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7) | 0 (0)
Cracks (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 8 (8) | 15 (15)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02751827/Prot_SAP_000.pdf